CLINICAL TRIAL: NCT03010241
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled Trial of Traditional Chinese Medicine in the Treatment of Diabetes Distal Symmetric Polyneuropathy
Brief Title: The Multi-Centric Clinical Study of Chinese Medicine Intervention on Diabetes Distal Symmetric Polyneuropathy.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Zhengzhou City Hospital of Traditional Chinese Medicine (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); Hebei Yiling Hospital (Other); Hubei Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lian-fengmei, PHD, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016Tangbi Prescription
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Distal Symmetric Polyneuropathy; Chinese medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Prescriptions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tangbi Prescription (Experimental): Based on the standard medical care, experimental group were treated with Tangbi Prescription 4.87g granules, 2 times/d, which The prescripton was composed by five Chinese herbal medicines.
  Interventions: Drug: Tangbi (prescription)
- Placebo (Placebo Comparator): Based on the standard medical care, placebo-controlled group were treated with Placebo 4.87g granules, 2 times/d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tangbi (prescription) — A kind of Granule(Tang bi fang) was made from five kind of Chinese herbs. Other: Standard medical care Standard medical care is in accordance with China Guideline for type 2 diabetes (2013).
  Other Names: Tang bi fang
  Arms: Tangbi Prescription
Drug: Placebo — Granule(Placebo) is in accordance with Tangbi prescription in appearance, colour, taste.
  Other: Standard medical care. Standard medical care is in accordance with China Guideline for type 2 diabetes (2013).
  Other Names: Placebos
  Arms: Placebo

SUMMARY:
Background: Distal symmetric polyneuropathy (DSPN) is the most common complication of type 2 diabetes mellitus (T2DM) and the most common form of peripheral neuropathy. DSPN increases the risk of foot ulceration up to seven-fold, and is a significant risk factor in more than 60% of the amputations of the lower limbs in patients with T2DM. Reportedly, TCM may have some advantages in relieving symptoms and reducing the incidence of DSPN exacerbations.We postulate that patients with DSPN will benefit from therapy with TCM treatment according to syndrome differentiation.

Methods and design: A randomized, double-blind, placebo-controlled and multi-centric clinical trial design was used on the basis of a co-regimen of mecobalamin. Subjects who met the inclusion criteria were randomly divided into two groups. The patients in the study group were treated with Tangbi prescription, and the patients in the control group were treated with placebo. Treatment was scheduled for 24 weeks. The sample size was 188 cases.Major evaluation indicators: Changes in Clinical Symptoms and Signs in Distal Symmetrical Polyneuropathy patients.The clinical symptoms and signs of patients were recorded by Michigan Diabetic Neuropathy Score(MDNS), and the changes of Michigan Diabetic Neuropathy Score(MDNS) were compared between the two groups before and after medication. Secondary Evaluation Indicators:① nerve conduction velocity changes, The changes in nerve conduction velocity of each nerve were compared before and after taking medicine.② Clinical symptoms and signs change, The clinical symptoms and signs of the patients were compared before and after taking the medicine.

Discussion: We postulate that patients with DSPN will benefit from therapy with TCM treatment.

DETAILED DESCRIPTION:
1. Purpose of the study Major objective: To evaluate the efficacy of traditional Chinese medicine (Tangbi prescription) in improving the clinical symptoms of patients with diabetic distal symmetric polyneuropathy.

   Secondary objective: To evaluate the effect of traditional Chinese medicine (Tangbi prescription) on nerve conduction velocity of patients with diabetic distal symmetric polyneuropathy.
2. Experimental Measures and contrast A randomized, double-blind, placebo-controlled and multi-centric clinical trial design was used on the basis of a co-regimen of mecobalamin. The patients in the study group were treated with Tangbi prescription (1 dose / day, twice), and patients were treated with placebo (1 dose / day, twice) in the control group. Treatment was scheduled for 24 weeks. The sample size was determined to 188 cases through statistics calculation.

   Sample size calculation basis: According to the preliminary study of Antang-tongbi prescription data, placebo group scale (Toronto TCSS scale) score difference is 3.45, while Tangbi prescription scale score was 4.14, and the public standard deviation s = 1.33. The sample size is estimated by hypothesis test formula of measurement data: N = 2 * [(Zα + Zβ) * δ / d] ^ 2 (pp. 112-113 of the third edition of Epidemiology) (n is the sample size and σ is the estimated standard deviation, d is two groups' continuous variable mean difference; Zα and Zβ are the corresponding standard normal differences; for Zα and Zβ values, see the Human Health Edition, Epidemiology, Third Edition, page 73, Table 6.2). Supposing= 0.05, β = 0.10, according to one-sided check table, the quantile Zα = 1.64485, Zβ = 0.84162, and put them into the formula, and result was n = 78.10. Therefore, each group needs 78 patients. Considering no more than 20% withdrawal rate, the total number of cases is 188, of 94 cases in each group.
3. Bias analysis The evaluation index of this study is clinical symptoms, affected by many factors. Although there are many ways in the treatment of oral drugs, but the exact evidence of evidence-based medicine is not proved. Therefore, there is little factor impacting of the biases of the evaluation results, concluding the following aspects: (1) blood glucose levels. (2) existing treatment measures, (3) the conditions of EMG determination.

   These influencing factors are addressed as follows: (1) As for blood glucose levels factor, a randomized, double-blind study design approach was used to ensure consistency of the factor in the two groups. (2) subjects taking Methycobal can reduce the psychological effect of patients on the efficacy of curative effect and increase patient compliance. (3) Train EMG doctors consistently, and the EMG determination is fixed, which forms the SOP of this study.
4. Research design 4.1 The design scheme A randomized, double-blind, placebo-controlled and multi-centric clinical trial design was used on the basis of a co-regimen of mecobalamin. Subjects who met the inclusion criteria were randomly divided into two groups. The patients in the study group were treated with Antang-tongbi prescription, and the patients in the control group were treated with placebo. Treatment was scheduled for 24 weeks. The sample size was 188 cases.

   4.2 Research Period Medication cycle is 24 weeks. 4.3 curative effect evaluation criteria 4.3.1 Major evaluation indicators Changes in Clinical Symptoms and Signs in Distal Symmetrical Polyneuropathy patients.

   The clinical symptoms and signs of patients were recorded by Michigan Diabetic Neuropathy Score(MDNS), and the changes of Michigan Diabetic Neuropathy Score(MDNS) were compared between the two groups before and after medication.

   4.3.2 Secondary Evaluation Indicators

   ① nerve conduction velocity changes The changes in nerve conduction velocity of each nerve were compared before and after taking medicine.

   ② Clinical symptoms and signs change The clinical symptoms and signs of the patients were compared before and after taking the medicine.

   4.4 Curative effect observation indicators ① Nerve conduction velocity (every 6 months).
   * MDNS scale (every 3 months). 4.5 Observational Indicators

     ① Background observation (0 weeks)
     1. Demographic data: gender, age, height, weight and so on.
     2. General clinical data: medical history, course of the disease, treatment history, combined disease and medication.
   * Diagnostic and monitoring indicators

     1. Blood pressure, fasting blood glucose test (every 1 month).
     2. Glycated hemoglobin, blood lipids (every 3 months). 4.6 Analysis of relevant measures are based on bias analysis 4.7 Basic treatment ① Diabetes education;
   * Diabetic diet;

     * Rational control of blood glucose: use oral hypoglycemic agents or insulin injections to keep all patients blood glucose stable in the study. In principle, the type and dose of hypoglycemic agents should maintain unchanged. If fasting blood glucose fluctuates more than 20%, diabetes experts were needed to find and remove the predisposing factors as soon as possible, and adjust the dose and monitor blood glucose changes, so the blood glucose can be smooth in 4 weeks. Adjusted dose of the drug needs to be detailed records in the combined medication table.

       ④ Taking Mecobalamin tablets (1 / time, 3 times / day). (Eisai (China) Pharmaceutical Co., Ltd.) 4.8 Provisions for combined treatment
       1. All Chinese herbal medicines with the same efficacy as the study drug (including Chinese herbal medicines with similar therapeutic indications and Chinese herbal medicines with similar efficacy) were banned during the study period.
       2. All combination therapy and treatment (treatment measure or treatment medicine of other diseases) should be documented in the combined medication table.
     * Besides Methycobal, drugs for the treatment of diabetic peripheral neuropathy are prohibited, including α-lipoic acid, epalrestat, VitB12 and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of diabetic distal symmetric polyneuropathy;
2. The patient's age is between 30-70 years;
3. Sign informed consent

Exclusion Criteria:

1. Recent use of antioxidants such as vitamin E or vitamin C, acute infection, liver and kidney dysfunction, acute complications of diabetes, severe cardiovascular and cerebrovascular diseases, neuropathy caused by long-term alcohol consumption and other factors.
2. Combined with cardiovascular, liver, kidney and hematopoietic system and other serious primary disease, serum transaminase beyond the normal value more than 2 times, serum creatinine greater than the upper limit of normal, psychiatric patients.
3. Pregnancy, prepared to pregnant or lactating women, or having a history of drug allergy.
4. Participate in other drug clinical within one month.
5. Systolic blood pressure> 160mmHg or diastolic blood pressure> 100mmHg.
6. Having the diabetic ketoacidosis, ketoacidosis and severe infection within one month.
7. Drinking alcohol excessive and/or taking psychoactive substances, drug abusers and dependents over the past five years.
8. Having other diseases or conditions may reduce the possibility of entry or complicate the entry according to the researchers' judgement, such as the working environment changes frequently, unstable living environment etc., what is easy to cause loss of contact.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-11 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
The clinical symptoms and signs of patients were recorded by Michigan Diabetic Neuropathy Score(MDNS), and the changes of Michigan Diabetic Neuropathy Score(MDNS) were compared between the two groups before and after medication | Month 0, Month 3, Month 6

SECONDARY OUTCOMES:
nerve conduction velocity changes The changes in nerve conduction velocity of each nerve were compared before and after taking medicine. | Month 0, Month 6
Clinical symptoms and signs change The clinical symptoms and signs of the patients were compared before and after taking the medicine. | Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jin D, Huang WJ, Meng X, Yang F, Zheng YJ, Bao Q, Zhang MZ, Yang YN, Ni Q, Lian FM, Tong XL. Chinese herbal medicine TangBi Formula treatment of patients with type 2 diabetic distal symmetric polyneuropathy disease: study protocol for a randomized controlled trial. Trials. 2017 Dec 29;18(1):631. doi: 10.1186/s13063-017-2345-1. PMID 29284520